CLINICAL TRIAL: NCT02243150
Title: First-In-Human Phase 1 Safety, Pharmacokinetic and Pharmacodynamic Study of G1T28-1 in Healthy Male and Female Subjects
Brief Title: Safety, Pharmacokinetic and Pharmacodynamic Study of the CDK 4/6 Inhibitor G1T28-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: G1T28-1-01
Record Dates: First submitted 2014-09-09; First posted 2014-09-17 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2015-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 (Experimental): 6mg/m2 of G1T28-1 or placebo will be administered in 50mL of 5% dextrose by IV infusion
  Interventions: Drug: G1T28-1 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 2 (Experimental): Dose of G1T28-1 or placebo will be determined based on the safety and PK data from Cohort 1; G1T28-1 or placebo will be administered in 50mL of 5% dextrose by IV infusion.
  Interventions: Drug: G1T28-1 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 3 (Experimental): Dose of G1T28-1 or placebo will be determined based on the safety and PK data from Cohort 2; G1T28-1 or placebo will be administered in 50mL of 5% dextrose by IV infusion.
  Interventions: Drug: G1T28-1 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 4 (Experimental): Dose of G1T28-1 or placebo will be determined based on the safety and PK data from Cohort 3; G1T28-1 or placebo will be administered in 50mL of 5% dextrose by IV infusion.
  Interventions: Drug: G1T28-1 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 5 (Experimental): Dose of G1T28-1 or placebo will be determined based on the safety and PK data from Cohort 4; G1T28-1 or placebo will be administered in 50mL of 5% dextrose by IV infusion. Subjects from this cohort may be selected to participate in the Whole Blood Ex-Vivo Stimulation group.
  Interventions: Drug: G1T28-1 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 6 (Experimental): Dose of G1T28-1 or placebo will be determined based on the safety and PK data from Cohort 5; G1T28-1 or placebo will be administered in 50mL of 5% dextrose by IV infusion. Subjects from this cohort may be selected to participate in the Whole Blood Ex-Vivo Stimulation group.
  Interventions: Drug: G1T28-1 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 7 - Bone Marrow Cohort (Experimental): All subjects in this cohort will receive active drug, G1T28-1. Dose of G1T28-1 will be determined based on the safety and PK data from previous cohorts. G1T28-1 will be administered in 50mL of 5% dextrose by IV infusion. Subjects in this cohort will be selected for the Ex-Vivo Stimulation group and will have a one time bone marrow aspirate at one of the following time points: pre dose, 12 or 24 hours post dose.
  Interventions: Drug: G1T28-1 (CDK 4/6 Inhibitor)

INTERVENTIONS:
Drug: G1T28-1 (CDK 4/6 Inhibitor)
Drug: Placebo
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6

SUMMARY:
This first-in-human (FIH) study will provide the first safety, PK, and PD data of G1T28-1 in humans and will allow further development of G1T28 1 in patients with cancer to reduce chemotherapy-induced myelosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18-60 years of age; no clinically significant findings reported following detailed physical examination, medical history, vital signs, clinical laboratory tests, and ECGs as deemed by the PI
* Body mass index (BMI) in the range of 18 to 32 kg/m2 (inclusive) and weighing at least 50 kg
* Non-smokers / non-users of nicotine containing products for at least the previous 3 months
* Agreement to use birth control during the study and 3 months post last visit
* Able to comply with all protocol requirements and procedures

Exclusion Criteria:

* Clinically significant abnormalities found during physical examination, medical history review, ECGs (including QTcf interval > 450 msec), vital signs and laboratory tests (including positive test for HIV, hepatitis B and/or C)
* History of any serious allergic reaction to any medication
* Participated in a previous clinical trial with an investigational product in the last 60 days
* Any blood or plasma donation or other loss of blood at a volume exceeding 500 mL within 3 months before dosing
* History of drug or alcohol abuse in the last 2 years and positive test for drug abuse
* Use of any systemic medication within the past 2 weeks, including use of herbal products
* Pregnant or lactating women
* Any other issue which, in the opinion of the PI, will make the subject ineligible for study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to day 14
  All Adverse events, including-clinical laboratory data, vital signs and ECGs will be analyzed in all subjects receiving study drug through 14 days post dose of study drug.

SECONDARY OUTCOMES:
Pharmacokinetics of G1T28-1 in Plasma: Peak Plasma Concentration (Cmax) | Day 1, Day 2, Day 3 and Day 4
  The observed peak plasma concentration determined from the plasma concentration vs. time data
Pharmacokinetics of G1T28-1 in Plasma: Time to reach the observed peak plasma concentration (tmax) | Day 1, Day 2, Day 3 and Day 4
  The time to reach the observed peak plasma concentration from the plasma concentration vs. time data
Pharmacokinetics of G1T28-1 in Plasma: Area under the plasma concentration -time curve from 0-12 hrs (AUC 0-12) | Day 1
  Area under the plasma concentration-time curve from 0 to 12 hours post dosing, calculated by linear/log trapezoidal method
Pharmacokinetics of G1T28-1 in Plasma: Area under the plasma concentration- time curve from 0 to last (AUC 0-last) | Day 1, Day 2, Day 3, Day 4
  Area under the plasma concentration-time curve from time 0 to time of last measurable concentration calculated by linear/log trapezoidal method
Pharmacokinetics of G1T28-1 in Plasma: Area under the plasma concentration-time curve from time zero to infinity | Day 1, Day 2, Day 3, Day 4
  Area under the concentration time curve from time zero extrapolated to infinity
Pharmacokinetics of G1T28-1 in Plasma: terminal half life (T1/2) | Day 1
  Terminal half-life, defined as 0.693 divided by λzλ
Pharmacokinetics of G1T28-1 in Plasma: Terminal phase rate constant | Day 1
  Determined by linear regression of at least 3 points on the terminal phase of the log-linear plasma concentration-time curve.
Pharmacokinetics of G1T28-1 in Plasma: Clearance | Day 1
  Clearance after intravenous administration
Pharmacokinetics of G1T28-1 in Plasma: Volume of distribution | Day 1
  Volume of distribution in the terminal elimination phase
Pharmacodynamics-Whole Blood Ex Vivo Stimulation | Day 1
  Analysis of peripheral blood cell proliferation
Pharmacodynamic - Bone Marrow Analysis | Day 1
  Analysis of hematopoietic stem and progenitor cell (HSPC)

CONTACTS AND LOCATIONS:
Overall Officials: Renger Tiessen, MD, Principal Investigator — PRA Clinic Netherlands
Locations (1):
- PRA Early Development Clinic, Groningen, Netherlands

REFERENCES:
- [Derived] Li C, Hart L, Owonikoko TK, Aljumaily R, Rocha Lima CM, Conkling PR, Webb RT, Jotte RM, Schuster S, Edenfield WJ, Smith DA, Sale M, Roberts PJ, Malik RK, Sorrentino JA. Trilaciclib dose selection: an integrated pharmacokinetic and pharmacodynamic analysis of preclinical data and Phase Ib/IIa studies in patients with extensive-stage small cell lung cancer. Cancer Chemother Pharmacol. 2021 May;87(5):689-700. doi: 10.1007/s00280-021-04239-9. Epub 2021 Feb 17. PMID 33595690